CLINICAL TRIAL: NCT02762565
Title: Clinical Utility of a Low-Cost Hand-Held Breast Scanner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: UPCC 24114
Record Dates: First submitted 2016-04-25; First posted 2016-05-05 (Estimated); Results first posted 2021-04-29 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-05

CONDITIONS: Symptomatic Breast Lump

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- breast scanner (Experimental)
  Interventions: Device: PEFS system (Product Name: Intelligent Breast Exam™ or iBE™

INTERVENTIONS:
Device: PEFS system (Product Name: Intelligent Breast Exam™ or iBE™

SUMMARY:
Early detection of breast cancer improves the survival rate and makes treatment less costly. This study would measure the accuracy a low-cost hand-held commercially viable device, iBE, for the detection of clinically relevant findings in the breast using the results of current mammography as a comparison. This research will have no impact on clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Women and men with symptomatic breast lump (either by palpation or imaging) OR
* Asymptomatic women presenting to the imaging center for a screening mammogram.
* Signed Informed Consent

Exclusion Criteria:

* Patients under 18 years of age
* Patients who previously participated in this study and are returning to the Women's Imaging Center for follow-up diagnostic tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Brooks, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Breast Scanner: One time use of PEFS system (Product Name: Intelligent Breast Exam™ or iBE™) on breast
Period: Overall Study
Arm/Group | Breast Scanner
Started | 89
Completed | 78
Not Completed | 11
Not completed — Missing iBE data: a result of incomplete data transfer from the iBE | 11

BASELINE CHARACTERISTICS:
Population: 78 participants breast scanner information was complete transferred from the iBE device
Groups:
- Breast Scanner: PEFS system (Product Name: Intelligent Breast Exam™ or iBE™
Arm/Group | Breast Scanner
Number analyzed (Participants) | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 42 [21 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 69
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 27
  White | 44
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Quadrants With Detected Breast Lesions
Description: The iBE results were evaluated by definitive quadrants. The definitive quadrants break down the superimposed clock into 4 equal sectors (e.g. 12-3, 3-6, 6-9, 9-12).
Time Frame: 3 months
Population: the iBE result of each participant was broken into 4 quadrants for each breast. Some quadrants were missing iBE data. 78 participants and 342 quadrants, 77 is the number of quadrants with positive findings of the 78 participants and the 342 quadrants analyzed.
Measure: Count of Units; unit: quadrants
Units Other Than Participants: quadrants
Arm/Group | Breast Scanner
Number analyzed (Participants) | 78
Number analyzed (quadrants) | 342
quadrants
  Number of quadrants positive for a lesion | 77
  Number of quadrants negative for a lesion | 265

2. Primary Outcome: Sensitivity of iBE Breast Lesion Detection
Description: the number of quadrants with positive breast lesion detected by iBE confirmed by mammogram and ultrasound, 4 quadrants per breast per participant. 77 quadrants were labeled positive for breast lesion by iBE, 66 were confirmed positive by mammogram or ultrasound allowing calculation of sensitivity of the the iBE breast lesion detection
Time Frame: 1 day
Population: quadrants with positive breast lesions
Measure: Count of Units; unit: quadrants
Units Other Than Participants: quadrants
Arm/Group | Breast Scanner
Number analyzed (Participants) | 78
Number analyzed (quadrants) | 77
quadrants | 66

3. Primary Outcome: Specificity of iBE Breast Lesion Detection
Description: the number of quadrants characterized normal breast by iBE confirmed by mammogram and ultrasound, 4 quadrants per breast per participant
Time Frame: 1 day
Population: breast quadrants negative for breast lesions
Measure: Count of Units; unit: quadrants
Units Other Than Participants: quadrants
Arm/Group | Breast Scanner
Number analyzed (Participants) | 78
Number analyzed (quadrants) | 265
quadrants | 237

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Breast Scanner
All-Cause Mortality (participants affected / at risk) | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes